CLINICAL TRIAL: NCT00945282
Title: A Proof of Concept Study for GSK2248761 (An Extension of NV-05A-002: A Phase I/IIa Double-Blind Study to Evaluate the Safety and Tolerability, Antiretroviral Activity, Pharmacokinetics and Pharmacodynamics of IDX12899 in Antiretroviral Treatment-Naive HIV-1 Infected Subjects, Completed by Idenix)
Brief Title: Safety and Tolerability Study to Evaluate Lower Dose of GSK2248761 in Antiretroviral Treatment-Naive HIV-1 Infected Adults.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113020
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: IDX12899; adaptive; monotherapy; pharmacokinetics; Treatment-naive; HIV-1; GSK2248761; NNRTI; HIV Infections; treatment naive
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — IDX 899; Lopinavir; lopinavir-ritonavir drug combination; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): In Cohort 1 subjects will receive either GSK2248761 30 mg or placebo once a day for 7 days. On Day 8 subjects will receive either Kaletra or HAART for 28 days. The doctor will choose the most appropriate medications for HAART.
  Interventions: Drug: GSK2248761; Drug: Lopinavir/ritonavir; Drug: HAART; Drug: Placebo
- Cohort 2 (Experimental): In Cohort 2 subjects will receive either GSK2248761 in the range of 10 mg - 20 mg or 40 mg - 90 mg or placebo once a day for 7 days. On Day 8 subjects will receive either Kaletra or HAART for 28 days. The doctor will choose the most appropriate medications for HAART. The dose for Cohort 2 will be determined following evaluation of results from Cohort 1. Cohort 2 may not be done.
  Interventions: Drug: Lopinavir/ritonavir; Drug: HAART; Drug: Placebo; Drug: GSK2248761

INTERVENTIONS:
Drug: GSK2248761 — GSK2248761 30 mg capsule once a day for 7 days. GSK2248761 is an investigational (not approved by the FDA) HIV drug in the class of non-nucleoside reuptake inhibitor class.
  Arms: Cohort 1
Drug: Lopinavir/ritonavir — Lopinavir 400 mg and ritonovir 100 mg every 12 hours for 28 days. Lopinavir/ritonavir is approved by the FDA as an HIV medication in the protease inhibitor class. Kaletra is a trademark of Abbott Laboratories.
  Other Names: Kaletra
Drug: HAART — Highly Active Antiretroviral therapy of the doctor's choice.
Drug: Placebo — Placebo is a capsule with no drug in it.
Drug: GSK2248761 — GSK2248761 10 mg -20 mg or 40 mg - 90 mg once a day for 7 days. GSK2248761 is an investigational (not approved by the FDA) HIV drug in the class of non-nucleoside reuptake inhibitor class.
  Arms: Cohort 2

SUMMARY:
GSK has in-licensed a novel NNRTI-class candidate (GSK2248761, IDX12899) for the treatment of subjects with HIV-1 infection from Idenix Pharmaceuticals. Idenix Pharmaceuticals completed a proof-of-concept study evaluating GSK2248761 monotherapy over seven days in forty treatment-naïve subjects infected with HIV-1. GSK2248761 doses sequentially evaluated were 800 mg QD, 400 mg QD, 200 mg QD and 100mg QD.

This study will evaluate a lower dose, or doses, of GSK2248761 to better characterize the dose-response and concentration-response curves. The results from this study will be used to select doses for future clinical studies in HIV-1 infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 21 to 65 years of age.
* Female of non-childbearing potential defined as: being post-menopausal, defined as 12 months of spontaneous amenorrhea and having a serum FSH level >40 MIU/ml at Screening OR have had a documented bilateral tubal ligation or hysterectomy of at least 6 months prior to study initiation, bilateral oophorectomy or bilateral tubal ligation.
* Plasma HIV-1 RNA value >= 5000 copies/mL.
* CD4+ count >= 200 cells/mm3.
* Is antiretroviral treatment-naïve and agrees not to start antiretroviral therapy prior to clinic check-in (Day-1).
* Subject agrees to start a standard HAART regimen on Day 8 of the study or Kaletra monotherapy for 28 days within 24 hours after the last dose of study medication.
* Capable of giving written informed consent, which includes being willing and able to comply with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subject is pregnant as determined by a positive urine/serum pregnancy test at Screening and Day -1.
* Lactating females.
* Male subjects of reproductive potential and unwilling to use double barrier method of contraception (e.g., condom plus spermicide) and continue to use an adequate method of birth control for at least 30 days after the last dose of the study drug.
* Has a positive screening Hepatitis B surface antigen, positive screening Hepatitis C virus (HCV) antibody and detectable HCV ribonucleic acid (RNA) on subsequent testing. If the Hepatitis C antibody is positive but the HCV RNA is undetectable, the subject may be included in the study.
* History of regular alcohol consumption within 6 months of Screening as defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits
* Has a positive pre-study drug screen. Drugs that will be screened for include amphetamines, barbiturates, cocaine and PCP.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the Principal Investigator, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.

Note: Study drugs include GSK2248761 placebo or the follow-up HAART or Kaletra therapy.

* Received an immunomodulating agent (e.g., interleukin-2) or immunotherapeutic vaccine within 30 days before Day -1.
* Requires a medication that is a known substrate, inhibitor and/or inducer of CYP3A4.
* Has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dosing day.
* Has ever had an AIDS-defining illness.
* Has a history of or has a currently active clinically important disease other than HIV-1 infection that, in the opinion of the Investigator, may put the subject at risk because of participation in this study (including renal and hepatic impairment, active infections including tuberculosis or opportunistic infection, malignancy and cardiac dysfunction).
* Has an intestinal malabsorption (e.g., structural defects, digestive failure, enzyme deficiencies, etc).
* Has a pre-existing NNRTI drug resistance based on genotyping at Screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* Subject has any of the following laboratory parameters at Screening (a single repeat is allowed for eligibility determination): Hemoglobin <8.5 g/dL, Neutrophil count <1000 cells/mm3, Platelet count <100,000 cells/mm3, Serum creatinine > the upper limit of normal (ULN), AST or ALT <= 2.5 x ULN.
* Exclusion Criteria for Screening ECG (A single repeat is allowed for eligibility determination): Exclusion Criteria for Screening ECG: Heart rate: (males) <45 and >100 bpm (females) <50 and >100 bpm, QRS duration: >120 msec, QTc interval (Bazett): > 450 msec. Non-sustained (>= 3 consecutive beats) or sustained ventricular tachycardia. Sinus Pauses >2.5 seconds. 2nd degree (Type II) or higher AV block. Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization)).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10-20 (Actual); Primary Completion 2009-11-28 (Actual); Study Completion 2009-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buenos Aires, Argentina

REFERENCES:
- [Background] Zala C, St Clair M, Dudas K, Kim J, Lou Y, White S, Piscitelli S, Dumont E, Pietropaolo K, Zhou XJ, Mayers D. Safety and efficacy of GSK2248761, a next-generation nonnucleoside reverse transcriptase inhibitor, in treatment-naive HIV-1-infected subjects. Antimicrob Agents Chemother. 2012 May;56(5):2570-5. doi: 10.1128/AAC.05597-11. Epub 2012 Feb 6. PMID 22314532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants with Treatment-Naive, Human Immuno deficiency virus (HIV-1) infection were randomized to the study. The study was conducted from 20 October 2009 to 28 November 2009 at one center in Argentina.
Pre-assignment Details: One participant was initially enrolled in the study, however withdrew consent prior to randomization. The study was planned to be conducted in 2 cohorts, however based on safety and antiviral activity of Cohort 1, a second cohort of participants was not needed and the study was stopped.
Groups:
- GSK2248761 30 mg: Eligible participants received 3 capsules of GSK2248761 10 milligrams (mg) orally once daily dosed with 360 milliliter (mL) water after a standard breakfast, upto 7-days. Participants were to have fasted 4 hours after dosing. Unless otherwise instructed participants were not to recline (remained upright) for the first 4 hours following oral administration. On Day 8 participants received either Kaletra or Highly active antiretroviral therapy (HAART) for 28 days.
- Placebo: Eligible participants received matching placebo capsules to GSK2248761 10 mg capsules, orally once daily dosed with 360 mL water after a standard breakfast upto 7-days. Participants were to have fasted 4 hours after dosing. Unless otherwise instructed participants were not to recline (remained upright) for the first 4 hours following oral administration. On Day 8 participants received either Kaletra or HAART for 28 days.
Period: Overall Study
Arm/Group | GSK2248761 30 mg | Placebo
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2248761 30 mg: Eligible participants received 3 capsules of GSK2248761 10 mg orally once daily dosed with 360 mL water after a standard breakfast, upto 7-days. Participants were to have fasted 4 hours after dosing. Unless otherwise instructed participants were not to recline (remained upright) for the first 4 hours following oral administration. On Day 8 participants received either Kaletra or HAART for 28 days
- Placebo: Eligible participants matching placebo capsules to GSK2248761 10 mg capsules orally once daily dosed with 360 mL water after a standard breakfast upto 7-days. Participants were to have fasted 4 hours after dosing. Unless otherwise instructed participants were not to recline (remained upright) for the first 4 hours following oral administration. On Day 8 participants received either Kaletra or HAART for 28 days
- Total: Total of all reporting groups
Arm/Group | GSK2248761 30 mg | Placebo | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (7.10) | 28.0 (5.66) | 33.3 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, or is an important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or a drug-induced liver injury.
Time Frame: Up to 38 days
Population: Safety population was defined as all participants who were randomized into the study with documented evidence of receipt of at least one dose of randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Participants
  Any AE | 4 | 1
  Any SAE | 0 | 0

2. Primary Outcome: Change From Baseline in Hematology Paramaters- Basophils, Eosinophils, Lymphocytes, Monocytes, White Blood Cell Count
Description: The data for hematology parameters for Basophils, eosinophils, lymphocytes, monocytes, and white blood cell count from the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: thousand cells per microliter
Groups:
- GSK2248761 30 mg: Eligible participants received 3 capsules of GSK2248761 10 mg orally once daily dosed with 360 mL water after a standard breakfast, upto 7-days. Participants were to have fasted 4 hours after dosing. Unless otherwise instructed participants were not to recline (remained upright) for the first 4 hours following oral administration. On Day 8 participants received either Kaletra or HAART for 28 days. Eligible participants matching placebo capsules to GSK2248761 10 mg capsules orally once daily dosed with 360 mL water after a standard breakfast upto 7-days. Participants were to have fasted 4 hours after dosing. Unless otherwise instructed participants were not to recline (remained upright) for the first 4 hours following oral administration. On Day 8 participants received either Kaletra or HAART for 28 days.
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
thousand cells per microliter
  Basophils, Day 2 | -1.7 (4.08) | -5.0 (7.07)
  Basophils, Day 4 | 8.3 (9.83) | 5.0 (7.07)
  Basophils, Day 7 | 1.7 (7.53) | -10.0 (14.14)
  Basophils, Day 8 | 3.3 (8.16) | -10.0 (14.14)
  Basophils, Follow-Up | -3.3 (10.33) | -15.0 (7.07)
  Eosinophils, Day 2 | -1.7 (35.45) | -120.0 (141.42)
  Eosinophils, Day 4 | -60.0 (150.33) | -20.0 (0.00)
  Eosinophils, Day 7 | -38.3 (106.85) | -50.0 (28.28)
  Eosinophils, Day 8 | -96.7 (229.49) | -80.0 (70.71)
  Eosinophils, Follow-Up | -63.3 (153.84) | -135.0 (162.63)
  Lymphocytes, Day 2 | -120.0 (272.18) | 315.0 (1067.73)
  Lymphocytes, Day 4 | 268.3 (298.83) | 260.0 (296.98)
  Lymphocytes, Day 7 | 126.7 (415.44) | 180.0 (410.12)
  Lymphocytes, Day 8 | 273.3 (357.64) | 480.0 (1060.66)
  Lymphocytes, Follow-Up | -110.0 (375.34) | 50.0 (551.54)
  Monocytes, Day 2 | 28.3 (71.11) | 125.0 (176.78)
  Monocytes, Day 4 | 33.3 (76.59) | 120.0 (155.56)
  Monocytes, Day 7 | -15.0 (135.17) | 25.0 (77.78)
  Monocytes, Day 8 | 23.3 (103.67) | 75.0 (134.35)
  Monocytes, Follow-Up | 10.0 (143.67) | -115.0 (35.36)
  White blood cell, Day 2 | 148.3 (649.78) | 1295.0 (2849.64)
  White blood cell, Day 4 | 758.3 (896.78) | -10.0 (155.56)
  White blood cell, Day 7 | 45.0 (1017.70) | -600.0 (367.70)
  White blood cell, Day 8 | 500.0 (776.79) | -240.0 (1513.21)
  White blood cell, Follow-Up | -90.0 (699.29) | -110.0 (2573.87)

3. Primary Outcome: Change From Baseline in Hematology Paramaters- Hemoglobin
Description: The data for hematology parameter hemoglobin from the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: gram per decilitre
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
gram per decilitre
  Day 2 | -0.40 (0.316) | -0.50 (0.283)
  Day 4 | -0.28 (0.794) | 0.60 (1.273)
  Day 7 | -0.25 (0.864) | -0.45 (0.071)
  Day 8 | -0.48 (0.585) | -0.45 (0.354)
  Follow-up | -0.93 (0.550) | -1.00 (0.424)

4. Primary Outcome: Change From Baseline in Hematology Paramaters- Platelet Count
Description: The data for hematology parameter platelet count, for the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: per cubic millimeter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
per cubic millimeter
  Day 2 | -5.7 (24.86) | 3.0 (9.90)
  Day 4 | 5.0 (18.34) | -23.5 (37.48)
  Day 7 | 18.5 (19.77) | 2.5 (10.61)
  Day 8 | 29.3 (21.04) | 2.0 (2.83)
  Follow-up | 23.3 (6.50) | -1.0 (33.94)

5. Primary Outcome: Change From Baseline in Hematology Paramaters- Red Blood Cell Count
Description: The data for hematology parameter red blood cell count, for the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: million cells per microliter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
million cells per microliter
  Day 2 | -0.153 (0.1129) | -0.240 (0.0283)
  Day 4 | -0.112 (0.2601) | 0.200 (0.4525)
  Day 7 | -0.083 (0.2947) | -0.190 (0.0707)
  Day 8 | -0.170 (0.1764) | -0.170 (0.1556)
  Follow-up | -0.343 (0.2300) | -0.375 (0.1344)

6. Primary Outcome: Change From Baseline in Hematology Parameters- Total Neutrophil
Description: The data for hematology parameter total neutrophil count, for the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: giga cells per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
giga cells per liter
  Day 2 | 243.3 (499.83) | 980.0 (1753.62)
  Day 4 | 508.3 (692.05) | -375.0 (21.21)
  Day 7 | -30.0 (750.55) | -745.0 (49.50)
  Day 8 | 296.7 (535.82) | -705.0 (374.77)
  Follow-up | 76.7 (433.34) | 105.0 (2142.53)

7. Primary Outcome: Change From Baseline in Hematology Paramaters- Mean Corpuscle Hemoglobin (MCH)
Description: The data for hematology parameter MCH, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
picogram
  Day 2 | 0.07 (0.197) | 0.45 (0.495)
  Day 4 | 0.08 (0.147) | 0.05 (0.071)
  Day 7 | 0.03 (0.320) | 0.20 (0.283)
  Day 8 | 0.07 (0.151) | 0.10 (0.141)
  Follow-up | 0.13 (0.367) | 0.25 (0.071)

8. Primary Outcome: Change From Baseline in Hematology Paramaters- Mean Corpuscle Volume (MCV)
Description: The change from baseline data for hematology parameter MCV, was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
femtoliters
  Day 2 | 0.27 (1.109) | -0.10 (0.990)
  Day 4 | 0.15 (0.698) | -0.20 (0.990)
  Day 7 | -0.10 (0.341) | -0.40 (0.283)
  Day 8 | 0.13 (0.333) | -0.15 (0.354)
  Follow-up | 0.47 (0.753) | -0.50 (0.566)

9. Primary Outcome: Change From Baseline in Hematology Paramaters- Hematocrit
Description: The data for hematology parameter Hematocrit, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
percentage of red blood cells
  Day 2 | -1.22 (1.286) | -2.15 (0.212)
  Day 4 | -0.92 (2.110) | 1.70 (3.536)
  Day 7 | -0.80 (2.563) | -1.85 (0.495)
  Day 8 | -1.45 (1.508) | -1.55 (1.202)
  Follow-up | -2.78 (1.907) | -3.55 (0.919)

10. Primary Outcome: Change From Baseline in Hematology Paramaters-Mean Corpuscle Hemoglobin Concentration
Description: The data for hematology parameter Mean Corpuscle Hemoglobin concentration, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
percentage of red blood cells
  Day 2 | 0.02 (0.445) | 0.55 (0.778)
  Day 4 | 0.05 (0.373) | 0.15 (0.212)
  Day 7 | 0.07 (0.361) | 0.40 (0.283)
  Day 8 | 0.02 (0.214) | 0.15 (0.212)
  Follow-up | -0.03 (0.301) | 0.45 (0.212)

11. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters- Albumin and Total Protein
Description: The data for clinical chemistry parameters Albumin and total protein, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: gram per deciliter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
gram per deciliter
  Albumin, Day 2 | -0.17 (0.207) | -0.20 (0.000)
  Albumin, Day 4 | -0.08 (0.248) | 0.00 (0.000)
  Albumin, Day 7 | -0.10 (0.283) | -0.05 (0.212)
  Albumin, Day 8 | -0.05 (0.383) | -0.10 (0.000)
  Albumin, Follow-up | -0.07 (0.137) | 0.05 (0.071)
  Total protein, Day 2 | -0.45 (0.302) | -0.55 (0.212)
  Total protein, Day 4 | -0.10 (0.385) | -0.10 (0.283)
  Total protein, Day 7 | 0.10 (0.494) | 0.05 (0.071)
  Total protein, Day 8 | 0.00 (0.636) | -0.25 (0.071)
  Total protein, Follow-up | -0.30 (0.268) | -0.20 (0.283)

12. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Blood Urea Nitrogen, Triglycerides, Glucose, Creatinine, Calcium, Cholesterol, Total Bilirubin, and Direct Bilirubin.
Description: The data for clinical chemistry parameters- Blood urea nitrogen, triglycerides, glucose, creatinine, calcium, cholesterol, total bilirubin, and direct bilirubin. The change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
milligram per deciliter
  Blood urea nitrogen, Day 2 | 1.5 (7.20) | -1.0 (2.83)
  Blood urea nitrogen, Day 4 | 4.3 (5.32) | 4.0 (5.66)
  Blood urea nitrogen, Day 7 | 1.0 (7.67) | 3.5 (2.12)
  Blood urea nitrogen, Day 8 | 2.7 (6.38) | 5.5 (9.19)
  Blood urea nitrogen, Follow-up | -2.2 (7.41) | 1.0 (15.56)
  Triglycerides, Day 2 | -17.8 (19.05) | 5.0 (14.14)
  Triglycerides, Day 4 | -19.8 (16.47) | 5.5 (4.95)
  Triglycerides, Day 7 | 5.2 (21.44) | 20.5 (27.58)
  Triglycerides, Day 8 | 20.8 (63.05) | 34.0 (21.21)
  Triglycerides, Follow-up | -3.0 (12.63) | 114.0 (8.49)
  Glucose, Day 2 | 1.3 (9.18) | 6.0 (4.24)
  Glucose, Day 4 | 0.0 (10.92) | -0.5 (12.02)
  Glucose, Day 7 | -1.8 (7.86) | -1.0 (1.41)
  Glucose, Day 8 | -5.2 (10.72) | -5.0 (2.83)
  Glucose, Follow-up | 3.0 (5.76) | 10.0 (4.24)
  Creatinine, Day 2 | -0.048 (0.0770) | 0.000 (0.0000)
  Creatinine, Day 4 | 0.025 (0.0586) | 0.025 (0.0071)
  Creatinine, Day 7 | -0.003 (0.0455) | 0.035 (0.0919)
  Creatinine, Day 8 | -0.060 (0.0569) | -0.040 (0.1273)
  Creatinine, Follow-up | -0.003 (0.1183) | 0.060 (0.1273)
  Calcium, Day 2 | -0.25 (0.176) | -0.25 (0.071)
  Calcium, Day 4 | -0.13 (0.301) | 0.05 (0.071)
  Calcium, Day 7 | -0.40 (0.322) | -0.20 (0.141)
  Calcium, Day 8 | -0.47 (0.418) | -0.45 (0.354)
  Calcium, Follow-up | 0.08 (0.299) | 0.05 (0.071)
  Cholesterol, Day 2 | -11.8 (13.92) | -12.0 (8.49)
  Cholesterol, Day 4 | -15.3 (28.72) | -17.5 (10.61)
  Cholesterol, Day 7 | -12.0 (35.25) | -20.5 (7.78)
  Cholesterol, Day 8 | -8.3 (41.15) | -13.5 (0.71)
  Cholesterol, Follow-up | -5.5 (33.44) | -0.5 (17.68)
  Total bilirubin, Day 2 | -0.12 (0.160) | -0.10 (0.141)
  Total bilirubin, Day 4 | -0.08 (0.133) | -0.15 (0.071)
  Total bilirubin, Day 7 | -0.03 (0.121) | -0.05 (0.071)
  Total bilirubin, Day 8 | -0.08 (0.075) | -0.10 (0.000)
  Total bilirubin, Follow-up | 0.08 (0.240) | 0.00 (0.000)
  Direct bilirubin, Day 2 | -0.08 (0.041) | 0.00 (0.000)
  Direct bilirubin, Day 4 | -0.08 (0.041) | 0.00 (0.000)
  Direct bilirubin, Day 7 | -0.05 (0.055) | 0.05 (0.071)
  Direct bilirubin, Day 8 | -0.05 (0.055) | 0.00 (0.000)
  Direct bilirubin, Follow-up | 0.02 (0.075) | 0.10 (0.000)

13. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters- Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase
Description: The data for clinical chemistry paramaters- alkaline phosphatase, alanine amino transferase, aspartate amino transferase, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: International units (IU) per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
International units (IU) per liter
  Alkaline phosphatase, Day 2 | -5.8 (7.14) | -16.0 (0.00)
  Alkaline phosphatase, Day 4 | -1.5 (10.33) | -16.0 (8.49)
  Alkaline phosphatase, Day 7 | 1.8 (10.83) | -7.5 (4.95)
  Alkaline phosphatase, Day 8 | 3.3 (14.88) | -14.5 (6.36)
  Alkaline phosphatase, Follow-up | 4.2 (24.96) | -9.5 (0.71)
  Alanine amino transferase, Day 2 | -3.0 (6.63) | 0.5 (6.36)
  Alanine amino transferase, Day 4 | -2.0 (15.02) | -3.5 (4.95)
  Alanine amino transferase, Day 7 | 1.7 (21.81) | -3.5 (4.95)
  Alanine amino transferase, Day 8 | 3.7 (24.40) | 0.0 (5.66)
  Alanine amino transferase, Follow-up | -7.2 (21.81) | -1.5 (6.36)
  Aspartate amino transferase, Day 2 | 0.8 (4.17) | 1.0 (1.41)
  Aspartate amino transferase, Day 4 | -0.2 (7.31) | -4.5 (3.54)
  Aspartate amino transferase, Day 7 | -0.3 (7.69) | -3.0 (8.49)
  Aspartate amino transferase, Day 8 | 1.7 (9.40) | 0.0 (5.66)
  Aspartate amino transferase, Follow-up | -0.2 (8.40) | 2.5 (4.95)

14. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters-sodium, Potassium and Carbondioxide or Bicarbonate
Description: The data for clinical chemistry parameters- sodium, potassium and carbon dioxide or bicarbonate, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: milliequivalents per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
milliequivalents per liter
  Sodium, Day 2 | -1.2 (1.17) | -0.5 (2.12)
  Sodium, Day 4 | -0.8 (1.60) | 1.0 (1.41)
  Sodium, Day 7 | -1.5 (1.64) | 0.0 (0.00)
  Sodium, Day 8 | -1.7 (1.51) | -0.5 (0.71)
  Sodium, Follow-up | 2.3 (1.63) | 1.0 (1.41)
  Potassium, Day 2 | -0.02 (0.293) | -0.25 (0.071)
  Potassium, Day 4 | 0.10 (0.434) | 0.10 (0.566)
  Potassium, Day 7 | -0.17 (0.314) | -0.10 (0.000)
  Potassium, Day 8 | -0.18 (0.371) | -0.00 (0.141)
  Potassium, Follow-up | -0.08 (0.360) | -0.30 (0.424)
  Carbondioxide, Day 2 | -0.80 (2.384) | -1.35 (2.051)
  Carbondioxide, Day 4 | 3.17 (1.488) | 2.70 (4.101)
  Carbondioxide, Day 7 | 2.93 (1.850) | 3.60 (2.121)
  Carbondioxide, Day 8 | 0.87 (2.471) | 1.65 (1.768)
  Carbondioxide, Follow-up | 2.03 (2.187) | -0.30 (1.131)

15. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters- Phosphorus
Description: The data for clinical chemistry paramaters- phosphorous, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: millimole per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
millimole per liter
  Phosphorus, Day 2 | -0.05 (0.524) | -0.80 (0.707)
  Phosphorus, Day 4 | 0.07 (0.799) | 0.25 (0.212)
  Phosphorus, Day 7 | -0.17 (0.628) | -0.00 (0.141)
  Phosphorus, Day 8 | -0.27 (0.662) | -0.35 (0.071)
  Phosphorus, Follow-up | -0.58 (0.634) | -0.95 (0.071)

16. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters- Uric Acid
Description: The data for clinical chemistry parameters Uric acid, the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Micromole per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Micromole per liter
  Uric acid, Day 2 | 0.27 (0.250) | -0.55 (0.212)
  Uric acid, Day 4 | 0.17 (0.408) | -0.70 (0.283)
  Uric acid, Day 7 | -0.15 (0.561) | -0.80 (0.707)
  Uric acid, Day 8 | -0.60 (0.970) | -1.05 (0.071)
  Uric acid, Follow-up | -0.53 (0.784) | -0.80 (0.566)

17. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters- Thyroxine, Free
Description: The data for clinical chemistry parameters Thyroxine, free the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Picomole per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Picomole per liter
  Thyroxine free, Day 2 | -0.018 (0.0768) | 0.015 (0.0636)
  Thyroxine free, Day 4 | 0.108 (0.1320) | 0.190 (0.0283)
  Thyroxine free, Day 7 | 0.065 (0.1011) | 0.120 (0.1414)
  Thyroxine free, Day 8 | 0.117 (0.1221) | 0.130 (0.0424)
  Thyroxine free, Follow- up | 0.072 (0.1332) | 0.135 (0.1485)

18. Primary Outcome: Change From Baseline in Clinical Chemistry Paramaters- Thyroxine Total, Thyroxine Binding Globulin, Total T3.
Description: The data for clinical chemistry parameters Thyroxine total, thyroxine binding globulin, Total T3 the change from baseline was reported. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 2, 4 , 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Nanomoles per liter
  Thyroxine total, Day 2 | -0.60 (0.648) | -0.40 (0.707)
  Thyroxine total, Day 4 | -0.08 (0.979) | 0.50 (0.283)
  Thyroxine total, Day 7 | -0.28 (0.773) | 0.10 (0.707)
  Thyroxine total, Day 8 | 0.00 (0.874) | 0.00 (0.141)
  Thyroxine total, Follow-up | -0.37 (1.019) | 0.05 (1.202)
  Thyroxine binding globulin, Day 2 | -0.33 (5.645) | 2.00 (2.828)
  Thyroxine binding globulin, Day 4 | -5.00 (3.688) | -6.50 (3.536)
  Thyroxine binding globulin, Day 7 | -0.67 (7.005) | -3.00 (8.485)
  Thyroxine binding globulin, Day 8 | 0.17 (1.169) | -1.00 (2.828)
  Thyroxine binding globulin, Follow-up | -1.83 (2.787) | -1.00 (8.485)
  Total T3, Day 2 | -0.013 (0.1334) | 0.170 (0.2404)
  Total T3, Day 4 | 0.068 (0.2180) | 0.310 (0.2687)
  Total T3, Day 7 | -0.055 (0.1435) | 0.225 (0.2333)
  Total T3, Day 8 | -0.035 (0.1252) | 0.190 (0.0141)
  Total T3, Follow-up | -0.005 (0.1945) | 0.375 (0.1344)

19. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Triplicate 12-lead ECGs were collected at different timepoints, after participants were supine for 5 minutes, during the study using an ECG machine that automatically calculated the heart rate (HR) and measures PR, QRS, QT, and QTc intervals. The three consecutive determinations were collected 5 plus or minus 2 minutes apart and all three tracings were recorded. The participants with abnormal values categorized as abnormal clinically significant (CS) and not clinically significant (NCS) were reported.
Time Frame: Day 1, Day 4, Day 7, Day 8 and follow-up
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Participants
  Day 1, Pre-dose, NCS | 3 | 0
  Day 1, 4 hour, NCS | 2 | 0
  Day 1, 8 hour, NCS | 2 | 0
  Day 4, Pre-dose, NCS | 2 | 0
  Day 4, 4 hour, NCS | 2 | 0
  Day 4, 8 hour, NCS | 3 | 0
  Day 7, Pre-dose, NCS | 3 | 0
  Day 7, 4 hour, NCS | 3 | 0
  Day 7, 8 hour, NCS | 2 | 0
  Day 8, Pre-dose, NCS | 3 | 0
  Follow-up, NCS | 3 | 0

20. Primary Outcome: Change From Baseline in Vital Signs-systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital sign measurements for SBP and DBP after sitting for 5 minutes were measured. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 1, 4, 7 , Day 8 and Follow-up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
millimeters of mercury
  SBP, Day 1, 4 hour | 4.3 (6.35) | -4.5 (14.85)
  SBP, Day 4, Pre-dose | -0.7 (5.92) | 0.5 (17.68)
  SBP, Day 4, 4 hour | 3.0 (11.70) | 12.5 (14.85)
  SBP, Day 7, Pre-dose | 6.2 (6.94) | 6.5 (9.19)
  SBP, Day 7, 4 hour | 9.8 (2.71) | 14.5 (12.02)
  SBP, Day 8 | 8.5 (7.48) | 13.5 (19.09)
  SBP, Follow-up | 5.8 (7.33) | 14.5 (6.36)
  DBP, Day 1, 4 hour | 8.2 (8.16) | 1.0 (1.41)
  DBP, Day 4, Pre-dose | 5.8 (16.58) | 1.0 (15.56)
  DBP, Day 4, 4 hour | 9.7 (10.21) | 3.0 (12.73)
  DBP, Day 7, Pre-dose | 8.2 (10.96) | 7.0 (7.07)
  DBP, Day 7, 4 hour | 6.0 (9.80) | 8.0 (2.83)
  DBP, Day 8 | 5.2 (10.25) | 15.0 (9.90)
  DBP, Follow-up | 4.5 (9.07) | 8.0 (5.66)

21. Primary Outcome: Change From Baseline in HR
Description: Vital sign measurements for HR after sitting for 5 minutes were measured. The average mean values were measured. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose [Screening, Day -1 or Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose at Day -1 or Day 1) and Day 1 (4-hour), Day 4 (Pre-dose and 4 hour), Day 7 (pre-dose and 4-hour), Day 8 and follow up (Day 14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Beats per minute
  HR , Day 1, 4 hour | -2.5 (6.50) | -3.0 (4.24)
  HR, Day 4, Pre-dose | -2.7 (6.12) | -6.0 (11.31)
  HR, Day 4, 4 hour | -2.2 (3.92) | -6.0 (21.21)
  HR, Day 7, Pre-dose | 3.0 (7.54) | -1.0 (22.63)
  HR, Day 7, 4 hour | -0.3 (4.63) | -2.5 (17.68)
  HR, Day 8 | 3.7 (7.42) | 0.0 (12.73)
  HR, Follow-up | -0.3 (5.99) | 5.0 (11.31)

22. Primary Outcome: Change From Baseline Through Day 8 in Plasma HIV-1 RNA
Description: The quantitative analysis of plasma was done to evaluate the amount of HIV-1 RNA at Day 1,2,3,4,5,6,7, 8 and End of treatment visit. The quantification was done using a Polymerase chain reactor (PCR). The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose Day 1) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose Day 1) to Day 8
Population: The Intent-to-treat Exposed (ITT) Population was defined as all participants who met the study criteria and were randomized into the study with documented evidence of having received at least 1 dose of randomized treatment and at least one post-baseline HIV-1 RNA measurement and have Day 1 HIV-RNA>1500 copies/mL.
Measure: Mean (Standard Deviation); unit: log 10 copies per milliliter (mL)
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
log 10 copies per milliliter (mL) | -0.967 (0.3988) | -0.036 (0.2495)
Statistical Analysis 1: Comparison: GSK2248761 30 mg vs Placebo; Test type: Superiority; p = 0.042, ANCOVA; Mean Difference (Final Values) = -0.932, 95% CI 2-sided [-1.812 to -0.053]

23. Primary Outcome: Change From Baseline to Nadir in Plasma HIV-1 RNA
Description: The quantification of plasma HIV-1 RNA, was conducted for the change from baseline to on treatment nadir (maximum change) before starting HAART or Kaletra monotherapy on Day 8. The quantification was done using a PCR. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline (pre-dose Day 1]) was defined as last available scheduled assessment prior to time of the first dose unless it is specified otherwise.
Time Frame: Baseline (pre-dose Day 1) to Day 8
Population: ITT population.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
log10 copies/mL | -1.019 (0.3687) | -0.580 (0.0157)
Statistical Analysis 1: Comparison: GSK2248761 30 mg vs Placebo; Test type: Superiority; p = 0.221, ANCOVA; Mean Difference (Final Values) = -0.413, 95% CI 2-sided [-1.173 to 0.347]

24. Primary Outcome: HIV-1 Rate of Decline by Treatment
Description: The rate of decrease in the viral load of HIV-1 virus in response to individual treatment was measured. The viral load data was assumed to have a log normal prior distribution and followed linear decline with non-informative conjugate prior densities. The rate of decline (slope of the day) for each treatment was measured using a PCR from Day 1 to Day 8. The slope has been reported as mean.
Time Frame: Day 1 to Day 8
Population: ITT population.
Measure: Mean (90% Confidence Interval); unit: log10 copies/mL
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
log10 copies/mL | -0.1243 [-0.1478 to -0.1008] | 0.0189 [-0.0645 to 0.1023]
Statistical Analysis 1: Comparison: GSK2248761 30 mg; Day 1 to Day 8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The p-value is the value for GSK2248761 30 mg, at Day 1 to Day 8
Statistical Analysis 2: Comparison: Placebo; Placebo, Day 1 to Day 8; Test type: Superiority or Other; p = 0.6922, Mixed Models Analysis — The p-value is the value for placebo, at Day 1 to Day 8

25. Primary Outcome: GSK2248761 Pharmacokinetic (PK) Parameters Following Dose Administration on Day 1: Area Under the Plasma Concentration Time Curve 0 to Infinite (AUC[0-∞]) and Area Under the Plasma Concentration Time Curve (AUC [0-24])
Description: AUC (0-24), measured the plasma concentration of GSK2248761 against time, from time zero (pre-dose) to 24 hrs post-dose AUC (0-24) and from time zero to extrapolated infinite time AUC (0-∞). Serial blood samples were collected on Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 1 and used for analysis.
Time Frame: Day 1 (Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose)
Population: The PK Concentration Population included all participants who received GSK22648761 and underwent plasma PK sampling during the study. Participants for whom a plasma PK sample was obtained and assayed were included in the listing of plasma GSK2248761 concentration-time data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms (ng)/mL
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
hours*nanograms (ng)/mL
  AUC(0-inf) | 2217.73 (45)
  AUC(0-24) | 1842.19 (41)

26. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 1: Maximum Observed Concentration (Cmax) and Concentration at 24 Hours Post Dose (C24)
Description: Cmax represents the maximum concentration of GSK2248761 in the plasma. C24 is defined as the measure of plasma drug concentration of GSK2248761, 24 hours post dose, determined on Day 1. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 1 and used for analysis.Data for dose normalized Cmax and C24 was reported.
Time Frame: Day 1 (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours)
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
ng/mL
  Cmax | 585.43 (39)
  C24 | 103.40 (61)

27. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 7: Predose Concentration (C0), Concentration at End of Dosing Interval (Cτ), Minimum Observed Concentration During One Dosing Interval (Cmin) and Cmax
Description: The C0 was defined as the concentration of drug in plasma, before dose administration on Day 7. Cτ, was defined as the concentration of drug in the plasma at the end of dosing interval. The Cmin was defined as the minimum concentration of the drug in plasma during one dosing interval on Day 7. Cmax represents the maximum concentration of GSK2248761 in the plasma on Day 7. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 7 and used for analysis.
Time Frame: Day 7 (Pre -dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose)
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
ng/mL
  C0, Day 7 | 57.47 (83)
  Cτ, Day 7 | 54.27 (75)
  Cmin, Day 7 | 46.37 (83)
  Cmax, Day 7 | 212.93 (41)

28. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 1: Time to Maximum Observed Concentration (Tmax), Terminal Half-life (t1/2), Absorption Lag Time (Tlag)
Description: Tmax is defined as the, time of maximum measured GSK2248761 concentration in the plasma, on Day 1. The t1/2 was defined as the time measured for plasma concentration to decrease by one half. The tlag was defined as the time taken for the drug GSK2248761, to appear in the systemic circulation following administration. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 1 and used for analysis.
Time Frame: Day 1 (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose)
Population: PK population.
Measure: Median (Full Range); unit: hour
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
hour
  tmax | 4.00 [3.0 to 6.0]
  t1/2 | 7.99 [6.3 to 9.8]
  tlag | 0.49 [0.0 to 1.0]

29. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 1: Apparent Clearance (CL/F)
Description: The Clearance factor was defined as the volume of plasma cleared of the drug GSK2248761, per unit time. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 1 and used for analysis.
Time Frame: Day 1 (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose)
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
liter per hour | 13.53 (45)

30. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 7: AUC(0-τ)
Description: AUC(0-τ) is the AUC to the end of dosing period. For Day 7, it is the AUC measured at the end of the dosing period at Day 7. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 7 and used for analysis.
Time Frame: Day 7 (Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose)
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
hour*ng/mL | 9679.71 (54)

31. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 7: Tmax
Description: Tmax is defined as the, time of maximum measured GSK2248761 concentration in the plasma, on Day 7. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 7 and used for analysis
Time Frame: Day 7 (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose)
Population: PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
hours | 4.01 [3.0 to 6.0]

32. Primary Outcome: GSK2248761 PK Parameters Following Dose Administration on Day 7: t1/2
Description: The t1/2 was defined as the time measured for plasma concentration to decrease by one half. Serial blood samples were collected on Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 7 and used for analysis
Time Frame: Day 7 (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose)
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
hour | 9.69 (25)

33. Primary Outcome: Change From Baseline in CD4+ and CD8+ T-lymphocyte Cell Count at Day1 and Day 8.
Description: Whole venous blood samples were obtained from each participant for the analysis of lymphocyte subsets by flow cytometry (total lymphocyte counts, percentage, CD4+ cell counts, and CD8+ cell counts) at Screening, Day 1 and Day 8. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values (Day 1 and Day 8). Baseline was defined as Screening.
Time Frame: Baseline (Screening), Day 1 and Day 8
Population: ITT population.
Measure: Mean (Standard Deviation); unit: per cubic millimeter
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
per cubic millimeter
  CD4+ cells, Day 1 | 1.2 (76.32) | 76.0 (5.66)
  CD4+ cells, Day 8 | 87.5 (58.49) | 102.0 (107.48)
  CD8+ cells, Day 1 | 123.5 (348.90) | 526.0 (169.71)
  CD8+ cells, Day 8 | 313.3 (218.85) | 531.5 (539.52)

34. Secondary Outcome: Percent Change From Baseline in CD4+ and CD8+ T-lymphocyte Cell Count at Day 1 and Day 8
Description: Data for CD4+ and CD8+ cells was collected at Screening, Day 1 and Day 8. The percent change from baseline was reported at Day 1 and Day 8. Baseline was defined as Screening. The percent change from baseline was calculated as post-randomization value minus the baseline value.
Time Frame: Baseline (Screening), Day 1 and Day 8
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 6 | 2
Percent change
  CD4+, Day 1 | -3.2 (1.78) | -2.9 (1.27)
  CD4+, Day 8 | -2.4 (1.49) | -1.7 (0.42)
  CD8+, Day 1 | -2.8 (7.31) | 2.8 (3.82)
  CD8+, Day 8 | -0.4 (2.56) | 0.4 (1.41)

35. Secondary Outcome: Accumulation Ratio for AUC , Cmax, Cτ, and Time Invariance Ratio Following Repeat Administration
Description: The accumulation ratio is based on the parameters, Cmax, AUC(0-tau), AUC(0-24), C(tau), C24, AND AUC(0-inf). The accumulation ratio Ro was the ratio of AUC(0-tau) on Day 7 to that of AUC(0-24) on Day 1; the accumulation ratio R (Cmax) was the ratio of Cmax on Day 7 to that of Cmax on Day 1; the accumulation ratio R(Ctau) was the ratio of Ctau on Day 7 to the ratio of C24 on Day 1 and the Time Invariance Ratio Rs was defined as the ratio of AUC(0-tau) on Day 7 to that of AUC(0-inf) on Day 1. The ratio has been reported as number.
Time Frame: (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose ) on Day 1 and Day 7
Population: PK population.
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
ratio
  Accumulation Ratio Ro | 1.576 [1.321 to 1.880]
  Accumulation Ratio R [Cmax] | 1.212 [1.009 to 1.456]
  Accumulation Ratio R[Ctau] | 1.750 [1.170 to 2.617]
  Time Invariance Ratio Rs | 1.309 [1.094 to 1.567]

36. Secondary Outcome: Change From Baseline in Reverse Transcriptase Sequences of HIV-1 at Day 8
Description: None of the participants had non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance mutations at codons 90, 98, 100, 101, 103, 106, 108, 138, 179, 181, 188, 190, 225, or 230 at either Day 1 or Day 8. No mutation selected by GSK2248761 in vitro was observed for any participant at either Day 1 or Day 8. This data for "Change from baseline in reverse transcriptase sequences of HIV-1 at Day 8" not collected.
Time Frame: Baseline (Screening) and Day 8
Population: ITT population. Data not collected for "Change from baseline reverse transcriptase sequence"
Arm/Group | GSK2248761 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Assessment of the Achievement of Pre-dose GSK2248761 Steady State Concentration Following Repeat Dose Administration on Day 2 Through 7
Description: The pre-dose GSK2248761 steady state concentration, following repeated dose administration from Day 2 through Day 7 was assessed. Serial dose sampling was done on each day of Day 2, 3, 4, 5 and Day 6 and for Day 7 (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose), before the administration of the study drug daily.
Time Frame: Day 7 (Pre - dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose) and Days 2, 3, 4. 5 and 6: pre-dose only
Population: PK population.
Measure: Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | GSK2248761 30 mg
Number analyzed (Participants) | 6
ng/mL
  Days 4, 5, 6 and 7 | 0.052 [0.012 to 0.093]
  Days 5, 6 and 7 | -0.019 [-0.075 to 0.037]
  Days 6 and 7 | -0.056 [-0.230 to 0.118]

38. Secondary Outcome: PK Data of Day 1 AUC(0-inf) and Day 7 AUC(0-tau) at Different Doses for the Assessment of Dose Proportionality
Description: Data for IDX899 100 mg, IDX899 200 mg, IDX899 400 mg and IDX899 800 mg for Day 1 and Day 2 were taken from the Idenix NV-05A-002 study which were combined with GSK2248761 30 mg once daily data from this study, to assess the dose proportionality. The dose proportionality occurred when increase in the administered doses were accompanied by proportional increases in measure of exposure of the drug in the plasma PK parameters like AUC, Cmax, Ctau and other factors. The dose proportionality effects of IDX899 100 mg, IDX899 200 mg, IDX899 400 mg and IDX899 800 mg, following repeat dose administration on Day 7 for the PK parameter AUC(0-tau) has been reported.
Time Frame: (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose ) From Day 1 to Up to Day 7
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Groups:
- GSK2248761 30 mg: The eligible participants in this arm received GSK2248761 as 30 mg once daily for up to 7-days daily. On Day 8 participants received either Kaletra or HAART for 28 days.
- IDX899 100 mg: The eligible participants in this arm received IDX899 100 mg, once daily orally for upto 7-days daily. The dose was accompanied with 360 mL of water. On Day 8 participants received either Kaletra or HAART for 28 days. Data was taken from the Idenix NV-05A-002 study.
- IDX899 200 mg: The eligible participants in this arm received IDX899 200 mg, once daily orally for upto 7-days daily. The dose was accompanied with 360 mL of water . On Day 8 participants received either Kaletra or HAART for 28 days. Data was taken from the Idenix NV-05A-002 study.
- IDX899 400 mg: The eligible participants in this arm received IDX899 400 mg, once daily orally for upto 7-days daily. The dose was accompanied with 360 mL of water. On Day 8 participants received either Kaletra or HAART for 28 days. Data was taken from the Idenix NV-05A-002 study.
- IDX899 800 mg: The eligible participants in this arm received IDX899 800 mg, once daily orally for upto 7-days daily. The dose was accompanied with 360 mL of water. On Day 8 participants received either Kaletra or HAART for 28 days. Data was taken from the Idenix NV-05A-002 study.
Arm/Group | GSK2248761 30 mg | IDX899 100 mg | IDX899 200 mg | IDX899 400 mg | IDX899 800 mg
Number analyzed (Participants) | 6 | 8 | 8 | 8 | 8
hour*ng/mL
  AUC(0-inf), Day 1 | 2217.73 (45) | 9908 (21.07) | 23817 (46.77) | 33820 (58.30) | 37812 (81.37)
  AUC(0-tau), Day 7 | 2903.91 (54) | 11650 (31.02) | 27209 (47.46) | 49649 (26.55) | 53683 (72.34)

39. Secondary Outcome: PK Data of Cmax and Ctau at Different Doses for the Assessment of Dose Proportionality
Description: Data for IDX899 100 mg, IDX899 200 mg, IDX899 400 mg and IDX899 800 mg for Day 1 and Day 2 were taken from the Idenix NV-05A-002 study which were combined with GSK2248761 30 mg once daily data from this study, to assess the dose proportionality. The dose proportionality occurred when increase in the administered doses were accompanied by proportional increases in measure of exposure of the drug in the plasma PK parameters like AUC, Cmax, Ctau and other factors. Data for Ctau on Day 1 is presented for concentration at 24 hours post-dose on Day 1.
Time Frame: (Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose ) From Day 1 to Up to Day 7
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK2248761 30 mg | IDX899 100 mg | IDX899 200 mg | IDX899 400 mg | IDX899 800 mg
Number analyzed (Participants) | 6 | 8 | 8 | 8 | 8
ng/mL
  Cmax, Day 1 | 175.63 (39) | 797.8 (32.19) | 1686.2 (24.67) | 2625.9 (34.20) | 3406.4 (31.31)
  Cmax, Day 7 | 212.93 (41) | 960.1 (22.62) | 2158.9 (35.96) | 4140.7 (21.54) | 5394.5 (46.36)
  Ctau, Day 1 | 31.02 (61) | 128.9 (37.36) | 325.6 (60.93) | 422.9 (81.23) | 364.5 (123.77)
  Ctau, Day 7 | 54.27 (75) | 204.7 (48.36) | 469.2 (63.17) | 864.5 (47.44) | 540.3 (124.71)

ADVERSE EVENTS:
Time Frame: Up to 38 Days
Description: Safety population
Groups:
- GSK2248761 30 mg: The eligible participants in this arm received GSK2248761 as 30 mg once daily for up to 7-days daily . On Day 8 participants received either Kaletra or HAART for 28 days.
- Placebo: The eligible participants in this arm received matching placebo once daily for 7-days. On Day 8 participants received either Kaletra or HAART for 28 days
Arm/Group | GSK2248761 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 4/6 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2248761 30 mg (N=6) | Placebo (N=2)
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.